CLINICAL TRIAL: NCT03104673
Title: Molecular Signature of Karen and Burmese Children Until Two Years of Age on the Thailand--Myanmar Border: a Study Extension of TMEC 15-062
Brief Title: Molecular Signature Children
Acronym: MSP_Ext
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Sidra Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1502 Ext
Record Dates: First submitted 2017-03-08; First posted 2017-04-07 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Preterm Birth
Keywords: Molecular signature; Thailand-Myanmar border
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Early childhood Transcriptome from capillary blood (Risk-minimum) This point will enable us to understand whether preterm infants have different gene expression than their term counterparts and if so, how it evolves in the early period of life. Moreover, specific signals for children at risk for or suffering from malnutrition or stunting resulting from gastrointestinal inflammation or barrier disruption could be picked up. Total blood 0.85 mL in 2 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preterm birth (PTB) occurs before 37 weeks of gestation and is a major cause of neonatal mortality and morbidity. PTB results from heterogeneous influences. One of them is the inherited predisposition of spontaneous PTB, and another is the change in the placental microbial composition as this can cause infections, which lead to inflammation, a common cause of preterm birth. Interestingly, maternal periodontal disease is an independent risk factor for PTB, low birth weight and fetal growth restriction. Immune responses to infectious events or inflammation as well as genetic predisposition to inherited conditions have successfully been studied by using assessing genetic expression profiling. The molecular signature is sets of genes, proteins, genetic variants or other variables that can be used as markers for a particular phenotype.

Child morbidity from malnutrition resulting in poor growth and stunting remains a major public health issue that affects the local population just like PTB. While risk factors for malnutrition are multifaceted, there is also a hypothesized causal link between early gut microbiome disruption that leads to chronic malnutrition in otherwise healthy infants.

Molecular signatures including the intestinal microbiome development of preterm infants will be evaluated and compared to the term (≥37 weeks' gestation) counterparts. Moreover, a comprehensive examination of possible factors associated with poor growth and poor motor- and neurodevelopment will be assessed.

In this extension study: The primary goal for the child is to evaluate the perturbation in the development of the genomic profile including intestinal microbial habitat from children in a rural and limited-resource setting from birth to two years of life.

DETAILED DESCRIPTION:
Rationale:

The importance of early life epigenetics is now recognized to have direct implications for health in later life and a consistent limitation expressed in peer reviewed publications has been the small sample size of the studies. Rather than establish a separate cohort to study epigenetics in young children in this environment this extension study of TMEC 15-062 (Molecular signature of Karen and Burmese women on the Thailand--Myanmar border) aims to build on the detailed sampling of the mothers to not only identify biomarkers of preterm labor but also to understand high rates of stunting and anaemia in this area, and possibly develop predictive tools or pave new ways for prevention in the future.

Moreover, a non-invasive intervention in the form of nutrition and WASH counselling may provide information on whether this form of engagement can positively influence child development, prevent malnutrition and whether perturbations in the infants molecular signature can be observed.

In addition, the mothers exposed to the sampling procedure at birth in this study will be able to make a well-informed decision about whether they wish to enrol the child in such a study.

The rationale for the planned samples in children born to mothers who participated in the TMEC 15-062 study are summarized in the following text:

Child gut microbiome and assessment of nutrition from stool samples (Risk-none) The intestinal ecosystem is very dynamic, especially in the first period of life, as it needs to evolve from scratch, hence investigators want to follow children and analyse stool samples in first 24 month of life. investigators propose to assess what kind of impact the gut microbiome has on the child's growth and development. Since exposure to helminths is common in the study population, children stool samples will also be used to examine for helminthic infestations.

This point would also include a home visit as part of nutrition evaluation by questionnaire and direct observation (food preparation including hygiene, child food content, feeding patterns) to relate to microbiome.

Early childhood Transcriptome from capillary blood (Risk-minimum) This point will enable us to understand whether preterm infants have different gene expression than their term counterparts and if so, how it evolves in the early period of life. Moreover, specific signals for children at risk for or suffering from malnutrition or stunting resulting from gastrointestinal inflammation or barrier disruption could be picked up. Total blood 0.85 mL in 2 years.

Early childhood detection of anaemia from capillary blood (Risk-minimum) Anaemia will be treated and iron supplement effect on gut microbiome analysed. Total blood 0.85 mL in 2 years.

Early childhood detection of soil transmitted helminth infection from stool sample (Risk-none) Helminth infection will be treated and the effect on gut microbiome analysed. Stool sample each visit.

Child growth assessment and evaluation of motor and neurocognitive development (Risk-none) Premature infants have a higher risk for lifelong health and development problems. Investigators propose to follow the children's over the period of 2 years to assess their growth and their neurocognitive and motor development. Preterm children's growth and development will be compared to term neonates. The recommended schedule of growth assessment in healthy children is (1, 2, 4, 6, 9, 12, 18, 24 months). In this study children will be followed more frequently: monthly in the first year of life and 3 monthly in the 2nd year of life (1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 15, 18, 21, 24 months). The reasons for this include: the objective of the root study TMEC 15-062 which is on preterm infants who require closer follow up, to relate perturbations of biomarkers to stunting, and in this mobile population scheduled visits may be missed so a more flexible arrangement for checking anthropometry at any monthly visit in the first year of life reduces the chance that poor growth is not identified.

In addition, the growth and development of children born to mothers who had a febrile episode during pregnancy will be compared to children whose mothers did not experience fever episodes during pregnancy.

Children with poor growth or malnutrition will be given supplementary nutrition and nutrition advice will be given to the mother.

Grant reference number: B9R01250

ELIGIBILITY:
Inclusion Criteria:

* Karen or Burmese pregnant woman in study TMEC 15-062 who are willing to have their offspring (children) comply with all study requirements
* Pregnant woman is willing and able to give informed consent for her child to participate in this study

Exclusion Criteria:

* Children (in the investigators opinion) with any social or physical condition which would make it difficult to comply with study requirements

Inclusion Criteria for water, sanitation and hygiene (WASH) radomization

* Mother enrolled to MSP (TMEC 15-062) and child enrolled in MSP_Ext (TMEC 17-008)
* Term pregnancy (gestational age ≥37 weeks)
* Clinic birth
* Normal new-born
* Post-partum mother willing to have home visits
* Post-partum mother willing and able to give informed consent to participate in this study

Exclusion Criteria for water, sanitation and hygiene (WASH) randomization

* Lives too far to make home visits feasible
* Home situation unstable and likely to move before the child is 9 months old
* Social situation that would make it difficult for the mother to comply

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 400 children born from pregnant women who are attending antenatal care (ANC) clinics at Shoklo Malaria Research Unit and enrol into study TMEC 15-062. A subgroup of infants born to mothers with an uneventful pregnancy, normal vaginal clinic birth at term (estimated age of ≥ 37 weeks) will be approached and invited to participate in the randomised component of the trial.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Characterization of the molecular signature of child | at birth
  Early childhood Transcriptome from capillary blood
Characterization of the molecular signature of child | 1 year
  Early childhood Transcriptome from capillary blood
Characterization of the molecular signature of child | 2 years
  Early childhood Transcriptome from capillary blood
Proportions of nutrition and water, sanitation and hygiene (WASH) behaviours in home-based compared to clinic-based care | 9 months

SECONDARY OUTCOMES:
Proportion of children with biomarkers perturbations associated with poor child growth | From birth to two years of life.
  Describe the biomarkers predictive
Proportion of children with biomarkers perturbations associated with neurocognitive and motor development | From birth to two years of life.
  Describe the biomarkers predictive
Proportion of children with biomarkers perturbations associated with anaemia | From birth to two years of life.
  Describe the biomarkers predictive
Association between nutrition and water, sanitation and hygiene (WASH) behaviours and biomarker signature perturbations in children | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Tak, Mae Sot, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Volunteer's data and results from blood analyses stored in our database may be shared with other researchers to use in the future. However, the other researchers will not be given any information that could identify the subject.